CLINICAL TRIAL: NCT05195255
Title: Prebiotic Properties of Phenolic Compounds
Brief Title: Metabolic Response of Intestinal Microbiota to Guar Gum Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR(AG)33/2021B
Record Dates: First submitted 2021-11-11; First posted 2022-01-18 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: intestinal gas; healthy subjects; microbiota; prebiotic
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Prebiotic administration
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Guar gum (8 g/d) will be administered for 18 days

SUMMARY:
Some components of the diet are not absorbed in the small intestine and pass into the colon, where they may be fermented by the microbiota, releasing gas. A series of recent studies suggest that some non-absorbable, fermentable meal products (prebiotics) serve as substrate to colonic bacteria and change their composition, thereby producing beneficial effects to the host. These products are fermented by bacteria and at initial intake increase gas production; however, after 7-10 days administration some prebiotics induce an adaptation of intestinal microbiota towards more efficient metabolic pathways with less gas production. Hence, intestinal gas production may serve as an index of microbiota metabolic activity. Gas production may induce gas-related symptoms, such as flatulence, abdominal bloating and distention, and the symptoms improve when the microbiota adapts to the prebiotic and gas production declines. Guar gum is classified as a fiber, but it remains uncertain whether and to what extent it is fermented by colonic microbiota and whether it has prebiotic properties. Aim: to determine the metabolic reaction of intestinal microbiota in response to guar gum consumption, specifically, the extent of initial fermentation and subsequent adaptation.Design: Single-centre, single arm, open label, proof-of-concept study testing the effect of guar gum on microbiota metabolism and adaptation in healthy subjects Intervention: guar gum (8 g/d) will be administered for 18 days. Outcomes: during 4 days immediately before, at the beginning and at the end of the administration phase participants will be put on a standard diet and the following outcomes will be measured: a) number of gas evacuations during daytime for 2 days by means of an event marker; b) perception of digestive sensations by daily scales; c) microbiota composition by fecal analysis; d) metabolites in urine.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* gastrointestinal symptoms
* recent (3 months) antibiotic intake
* change in dietary habits 4 weeks before

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Number of daily anal gas evacuations | 18 days
  Change in the number of anal gas evacuations measured by an event marker from beginning of treatment to end of treatment

SECONDARY OUTCOMES:
Microbiota composition by fecal analysis | 18 days
  Change from beginning of treatment to end of treatment
Sensation of flatulence by scales | 18 days
  Sensation of flatulence measured on a 0-10 scale graded from 0 (no flatulence) to 10 (very intense sensation). Change from beginning of treatment to end of treatment
Sensation of abdominal bloating by scales | 18 days
  Sensation of abdominal bloating measured on a 0-10 scale graded from 0 (no bloating) to 10 (very intense sensation). Change from beginning of treatment to end of treatment.
Sensation of digestive well-being by scales | 18 days
  Sensation of digestive well-being measured on a -5 to +5 scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation). Change from beginning of treatment to end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain